CLINICAL TRIAL: NCT04065555
Title: Evaluation of TAK-981 and TAK-981 Combinations Following Intratumoral CIVO® Microdosing in Patients With Head and Neck Cancer
Brief Title: Intratumoral Microdosing of TAK-981 in Head and Neck Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Presage Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PBI-TAK-01
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Head and Neck Cancer
Keywords: precision oncology; intratumoral microdosing; microdose injection; microinjection; microdosing; in vivo oncology; in vivo drug sensitivity; tumor microenvironment; multiplexed immunohistochemistry; HNSCC; SCCHN
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — TAK-981; Cetuximab; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CIVO Microdose Injection of TAK-981, Cetuximab, and Avelumab (Experimental): Patients who are scheduled for surgical biopsy or tumor resection surgery will be injected one day (Cohort 1) or three days (Cohort 2) prior to surgery using the CIVO device. Each needle of the CIVO device will deliver up to 8.3 microliters of solution, including a vehicle control (sterile saline) or subtherapeutic microdoses of TAK-981, cetuximab, avelumab, TAK-981 combined with cetuximab, or TAK-981 combined with avelumab. Each microdose is simultaneously injected in a columnar fashion through each of 8, 5, or 3 needles (in a device configuration determined by tumor dimensions) into a single solid tumor or effaced metastatic lymph node. Approximately six patients will be assigned to each time point cohort. Cohort assignment is not sequential and will be selected by the Investigator based on clinic logistics and patient scheduling. Should one cohort fill in advance of the other, sites will be directed by Presage to enroll patients into the second cohort only.
  Interventions: Drug: TAK-981; Biological: Cetuximab; Biological: Avelumab; Combination Product: TAK-981 + Cetuximab; Combination Product: TAK-981 + Avelumab

INTERVENTIONS:
Drug: TAK-981 — Intratumoral microdose injection by the CIVO device.
Biological: Cetuximab — Intratumoral microdose injection by the CIVO device.
  Other Names: ERBITUX
Biological: Avelumab — Intratumoral microdose injection by the CIVO device.
  Other Names: Bavencio
Combination Product: TAK-981 + Cetuximab — Intratumoral microdose injection by the CIVO device.
  Other Names: TAK-981 + ERBITUX
Combination Product: TAK-981 + Avelumab — Intratumoral microdose injection by the CIVO device.
  Other Names: TAK-981 + Bavencio

SUMMARY:
This is a multi-center, single arm, open-label, multi-agent, localized pharmacodynamic biomarker Phase 0 trial designed to study the biological effects within the tumor microenvironment of TAK-981 and TAK-981 combined with cetuximab or avelumab when administered intratumorally in microdose quantities via the CIVO device. CIVO stands for comparative in vivo oncology.

DETAILED DESCRIPTION:
CIVO is a research tool composed of a hand-held single-use sterile injector coupled with fluorescent tracking microspheres called CIVO GLO that mark the sites of drug microdose injection, enabling rapid assessment of multiple oncology drugs or drug combinations simultaneously within a patient's tumor. In this Phase 0 intratumoral microdosing study in human patients with localized or metastatic primary tumors of the head and neck (who will be undergoing previously planned tumor and regional nodes dissection), we will evaluate TAK-981's ability to activate innate immune effector cells within the local tumor microenvironment. Additionally, this study will examine TAK-981 in combination with cetuximab or avelumab to study whether TAK-981 enhances the localized immune responses compared to those of either immunotherapy alone. TAK-981 singly and in combination with cetuximab or avelumab will be delivered intratumorally in subtherapeutic microdose quantities via CIVO.

The CIVO device penetrates solid tumors and delivers subtherapeutic microdoses of up to eight anti-cancer agents or combinations of anti-cancer agents co-injected with CIVO GLO into discrete regions of the tumor. At the time of the planned surgical intervention (one or three days after the CIVO microdose injection), the injected tumor tissue is then excised and tumor responses are assessed via histological staining of tumor cross-sections sampled perpendicular to each injection column. Co-injection with CIVO GLO enables identification of each injection site during resection as well as in tissues stained for analysis. Because the platform delivers microdose amounts of each test agent or combination directly into the patient's tumor tissue, hypotheses can be tested earlier in the drug development process, consistent with the goals of the 2006 FDA Exploratory IND Guidance for Industry.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to comply with the study's visit and assessment schedule.
2. Male or female ≥ 18 years of age at Visit 1 (Screening).
3. Pathologic diagnosis of primary cancers of the head and neck.
4. Ability and willingness to provide written informed consent. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
5. At least one lesion (primary tumor, recurrent tumor, or effaced metastatic lymph node) ≥ 2 cm in the shortest diameter that is surface accessible for CIVO injection that may be guided by ultrasound if appropriate and for which there is a planned surgical intervention. Treatment plan may include adjuvant radiation or chemotherapy and patients must have no medical contraindication to surgery.
6. ECOG (Eastern Cooperative Oncology Group) performance status of 0-2.
7. Female patients who:

   * Are postmenopausal for at least one year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice two effective methods of contraception, at the same time, from the time of signing of the informed consent through four months after the tumor injection procedure, OR agree to completely abstain from heterosexual intercourse.
   * Agree to refrain from donating ova during study participation.

Male patients, even if surgically sterile (i.e., status post-vasectomy), who:

* Agree to practice effective barrier contraception during the entire study treatment period through four months after the tumor injection procedure, OR
* Agree to completely abstain from heterosexual intercourse.
* Agree to refrain from donating sperm during study participation.

Exclusion Criteria:

1. Tumors or effaced nodes that are anticipated by the Investigator to lack a sufficient volume of viable tumor tissue (based on available pre-operative imaging, pre-injection ultrasound imaging, or pathology reports) for CIVO injection due to size, location, necrosis, cysts, excessive stroma, fibrosis, or treatment-induced tissue changes. Lesions that have received neoadjuvant radiation therapy may lack sufficient viable tumor tissue for CIVO injection procedures.
2. Patients who have received prior treatment with cetuximab or immune checkpoint inhibitors.
3. Female patients who are both lactating and breastfeeding or have a positive serum pregnancy during the screening period or a positive urine pregnancy test on Day 1 before the tumor injection procedure.
4. Any uncontrolled intercurrent illness, condition, serious medical or psychiatric illness, or circumstance that, in the opinion of the Investigator, could interfere with adherence to the study's procedures or requirements, or otherwise compromise the study's objectives.
5. Patients with uncontrolled autoimmune diseases requiring treatment.
6. Patients with human immunodeficiency virus/acquired immune deficiency syndrome (HIV/AIDS) with uncontrolled viral load and CD4 (Cluster of Differentiation 4) less than 200.
7. Patients that have received a live vaccine within 4 weeks of the baseline/screening visit.
8. Patients with a sensitivity to Captisol.
9. Use of any of the following ≤ 2 weeks prior to CIVO injection:

   1. Immunosuppressive drugs (e.g., calcineurin inhibitors)
   2. Biological response modifiers for autoimmune disease
   3. Systemic glucocorticoids: oral or parenteral corticosteroids at a dose ≥ 20 mg/day prednisone, or equivalent Note: physiologic replacement dosing of steroids (≤ 3mg/m2/d prednisone or equivalent), low-dose corticosteroids for dye allergies prior to staging scans or use in anti-emetic prophylaxis for patients undergoing chemotherapy, or topical steroids, are allowed
   4. Hematopoietic growth factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Quantification of Cell Death and Immune Cell Biomarkers by Immunohistochemistry (IHC) and In-Situ Hybridization (ISH) in Resected Tissue | 1 or 3 days after microdose injection
  Quantification of biomarker-positive and biomarker-negative cells will be performed within the tumor microenvironment around each of the injection sites of each resected patient sample by IHC and ISH. An aggregate analysis of this quantification may be done across patient samples to evaluate trends in tumor response. List of biomarkers evaluated may include biomarkers for cell death (e.g. cleaved caspase 3), T-cells (e.g. CD3, CD8/Granzyme B), and natural killer (NK) or myeloid cells (e.g. CD56/Granzyme B, CD86, CD68).

SECONDARY OUTCOMES:
Number of Patients with Adverse Events | Up to 28 days after microdose injection
  Relationship of AE to study drug or CIVO device will be determined using an AE Relatedness Grading System.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Presage Biosciences
Locations (6):
- United States (6):
  - University of Michigan, Ann Arbor, Michigan
  - Northwell Health (Lenox Hill), New York, New York
  - Northwell Health (Monter Cancer Center), North New Hyde Park, New York
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Portland VA, Portland, Oregon
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klinghoffer RA, Bahrami SB, Hatton BA, Frazier JP, Moreno-Gonzalez A, Strand AD, Kerwin WS, Casalini JR, Thirstrup DJ, You S, Morris SM, Watts KL, Veiseh M, Grenley MO, Tretyak I, Dey J, Carleton M, Beirne E, Pedro KD, Ditzler SH, Girard EJ, Deckwerth TL, Bertout JA, Meleo KA, Filvaroff EH, Chopra R, Press OW, Olson JM. A technology platform to assess multiple cancer agents simultaneously within a patient's tumor. Sci Transl Med. 2015 Apr 22;7(284):284ra58. doi: 10.1126/scitranslmed.aaa7489. PMID 25904742
- [Background] Frazier JP, Bertout JA, Kerwin WS, Moreno-Gonzalez A, Casalini JR, Grenley MO, Beirne E, Watts KL, Keener A, Thirstrup DJ, Tretyak I, Ditzler SH, Tripp CD, Choy K, Gillings S, Breit MN, Meleo KA, Rizzo V, Herrera CL, Perry JA, Amaravadi RK, Olson JM, Klinghoffer RA. Multidrug Analyses in Patients Distinguish Efficacious Cancer Agents Based on Both Tumor Cell Killing and Immunomodulation. Cancer Res. 2017 Jun 1;77(11):2869-2880. doi: 10.1158/0008-5472.CAN-17-0084. Epub 2017 Mar 31. PMID 28364003
- [Background] Dey J, Kerwin WS, Grenley MO, Casalini JR, Tretyak I, Ditzler SH, Thirstrup DJ, Frazier JP, Pierce DW, Carleton M, Klinghoffer RA. A Platform for Rapid, Quantitative Assessment of Multiple Drug Combinations Simultaneously in Solid Tumors In Vivo. PLoS One. 2016 Jun 30;11(6):e0158617. doi: 10.1371/journal.pone.0158617. eCollection 2016. PMID 27359113
- [Background] Moreno-Gonzalez A, Olson JM, Klinghoffer RA. Predicting responses to chemotherapy in the context that matters - the patient. Mol Cell Oncol. 2015 Jun 10;3(1):e1057315. doi: 10.1080/23723556.2015.1057315. eCollection 2016 Jan. PMID 27308571
- [Background] Gundle KR, Deutsch GB, Goodman HJ, Pollack SM, Thompson MJ, Davis JL, Lee MY, Ramirez DC, Kerwin W, Bertout JA, Grenley MO, Sottero KHW, Beirne E, Frazier J, Dey J, Ellison M, Klinghoffer RA, Maki RG. Multiplexed Evaluation of Microdosed Antineoplastic Agents In Situ in the Tumor Microenvironment of Patients with Soft Tissue Sarcoma. Clin Cancer Res. 2020 Aug 1;26(15):3958-3968. doi: 10.1158/1078-0432.CCR-20-0614. Epub 2020 Apr 16. PMID 32299817
- See also: Presage Website — https://presagebio.com/